CLINICAL TRIAL: NCT04461106
Title: A Two-Phase Study to Investigate Novel Biomarkers of Egg Consumption and Social Marketing Effectiveness of Egg Hubs for Malawian Infants
Brief Title: A New Measure of Egg Consumption and the Effect of Social Marketing Eggs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter, Malawi (Unknown); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202007077
Record Dates: First submitted 2020-06-22; First posted 2020-07-08 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Nutritional Stunting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Marketing Campaign (Active Comparator): Select egg hubs will receive social marketing campaign which aims to raise awareness about the benefits of eggs - 'why eggs': increasing the value of eggs from a consumer perspective and encourage consumption of eggs by children (<5yrs) and pregnant/lactating women.
  Interventions: Other: Social Marketing Campaign
- No Social Marketing Campaign (No Intervention): Other egg hugs will not receive social marketing campaign.

INTERVENTIONS:
Other: Social Marketing Campaign — aims to raise awareness about the benefits of eggs - 'why eggs': increasing the value of eggs from a consumer perspective and encourage consumption of eggs by children (<5yrs) and pregnant/lactating women
  Arms: Social Marketing Campaign

SUMMARY:
About 1600 children 6 to 24 months old will be enrolled from 8 egg hubs. 4 hubs will be receive social marketing campaign to raise awareness about the benefits of eggs while the other 4 will not receive social marketing campaign. Children will provide a urine sample for analysis of metabolites to correlate with egg consumption.

ELIGIBILITY:
Inclusion Criteria:

* Health children between 6 and 24 months of age

Exclusion Criteria:

* acute malnutrition
* congenital abnormalities
* chronic debilitation disease such as heart disease, cerebral palsy, or HIV infection

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 815 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Amount of egg consumed daily | 12 Months
  As determined by urinary metabolite concentrations. The specific metabolites will be identified in the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Project Peanut Butter, Blantyre, Malawi

REFERENCES:
- [Background] Garcia-Perez I, Posma JM, Gibson R, Chambers ES, Hansen TH, Vestergaard H, Hansen T, Beckmann M, Pedersen O, Elliott P, Stamler J, Nicholson JK, Draper J, Mathers JC, Holmes E, Frost G. Objective assessment of dietary patterns by use of metabolic phenotyping: a randomised, controlled, crossover trial. Lancet Diabetes Endocrinol. 2017 Mar;5(3):184-195. doi: 10.1016/S2213-8587(16)30419-3. Epub 2017 Jan 13. PMID 28089709
- [Background] S C Sri Harsha P, Abdul Wahab R, Cuparencu C, Dragsted LO, Brennan L. A Metabolomics Approach to the Identification of Urinary Biomarkers of Pea Intake. Nutrients. 2018 Dec 4;10(12):1911. doi: 10.3390/nu10121911. PMID 30518059
- [Background] Koppmair S, Kassie M, Qaim M. Farm production, market access and dietary diversity in Malawi. Public Health Nutr. 2017 Feb;20(2):325-335. doi: 10.1017/S1368980016002135. Epub 2016 Sep 9. PMID 27609557
- [Background] Eaton JC, Rothpletz-Puglia P, Dreker MR, Iannotti L, Lutter C, Kaganda J, Rayco-Solon P. Effectiveness of provision of animal-source foods for supporting optimal growth and development in children 6 to 59 months of age. Cochrane Database Syst Rev. 2019 Feb 19;2(2):CD012818. doi: 10.1002/14651858.CD012818.pub2. PMID 30779870

DOCUMENTS (1):
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT04461106/ICF_000.pdf